CLINICAL TRIAL: NCT01750541
Title: Haloperidol vs. Valproate in the Management of Agitated Patients Presenting to the Emergency Department: A Randomized Clinical Trial
Brief Title: Haloperidol vs. Valproate in Agitation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Kamran Heydari, Assistant Professor of Emergency Medicine, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB-021; MOH-021 (Other: The Ministry of Health and Medical Education (MOHME))
Record Dates: First submitted 2012-12-07; First posted 2012-12-17 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Psychomotor Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Haloperidol; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Haloperidol (Active Comparator): Haloperidol 5mg intramuscular injection
  Interventions: Drug: Haloperidol
- Valproate (Active Comparator): Valproate single Infusion; 400 mg (weigh<60 kg), 500 mg (weight>60 Kg)
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Haloperidol
  Other Names: Haldol
  Arms: Haloperidol
Drug: Valproate
  Other Names: Depakene
  Arms: Valproate

SUMMARY:
The aim of this study is to compare the efficacy of haloperidol and valproate in management of people with agitation in emergency department

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psychomotor agitation
* aged 18 to 65 years

Exclusion Criteria:

* Pregnant patients
* Severe liver disease
* History of drug (haloperidol/valproate) allergy
* Readily amendable causes for the agitation (hypoxemia or hypoglycemia)
* Hypotension (systolic blood pressure (SBP) ≤ 90 mm Hg)
* Known history of liver disease or uncontrolled diabetes
* Noticeable or suspected head trauma
* Previous history of neuroleptic malignant syndrome
* Receiving psychotropic medication, neuroleptic agents or cholinesterase inhibitors at the time of enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Agitated Behavior Scale (ABS) score | within the first 30 minutes of treatment onset
  Patients were rated before medication administration and within 30 minutes afterwards according to Agitated Behavior Scale (ABS) score. Any statistically significant change in ABS score consider as positive effect of either intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Heydari, MD, Principal Investigator — Department of Emergency Medicine, Imam Hossein Hospital, Shahid Beheshti University of Medical Sciences, Tehran, Iran.
Locations (1):
- Department of Emergency Medicine, Imam Hossein Hospital, Tehran, Tehran Province, Iran